CLINICAL TRIAL: NCT05123001
Title: Wearable Sensors and Molecular Omics to Detect and Mitigate Cell Therapy Adverse Events
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Surbhi Sidana, MD, Associate Professor of Medicine (Blood and Marrow Transplantation and Cellular Therapy), Stanford University
Other Study IDs: IRB-60459; NCI-2022-00603 (Registry Identifier: National Cancer Institute: Clinical Trials Reporting Program)
Record Dates: First submitted 2021-10-29; First posted 2021-11-17 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hodgkin Lymphoma; Non Hodgkin Lymphoma; Leukemia; Multiple Myeloma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CAR-T patients monitored with wearable devices and microsampling: All participants will receive wearable sensors, provide blood microsamples, and use the Biostrap mobile app for data capture. These are observational data collection tools applied to the entire cohort.

SUMMARY:
The purpose of this study is to monitor physiological and molecular changes during and following CAR-T cancer cell therapy, towards improved management of adverse events including Cytokine Release Syndrome and neurotoxicity.

Our study aims are to improved early detection and precise management of adverse events for patients receiving Chimeric antigen receptor T- cell (CAR-T):

1. To assess the feasibility, including accuracy, usability, and usefulness of wearable sensors in CAR-T patients.
2. To generate comprehensive multiomic profile analysis following CAR-T therapy.
3. To perform integrated analysis of wearables sensor data, omics data, and symptom/clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be in the process of undergoing cancer cell therapy at Stanford University.

  * Adults > 18 years
  * Any cell target may be used. (e.g. CD19, CD22, Bispecific CD19/22, Bispecific CD19/20, etc.)
  * English speaking
  * Assessed ability for caregiver/patient to use wearable devices and independently perform blood microsample collection

Exclusion Criteria:

* In the investigator's judgment, the subject is unlikely to comply with all protocolrequired study visits or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) receiving standard-of-care CAR-T cell therapy at Stanford University. Participants must be English-speaking and able, with caregiver assistance, to use wearable monitoring devices and perform blood microsampling. Up to 15 patients will be enrolled in this pilot study.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Monitoring heart rate data | 28 days
  Defined as ≥70% of patients able to wear at least one sensor device for ≥50% of the days from CAR-T infusion (Day 0) to Day 28.
  Each day is counted if ≥12 hours of data are captured.
Monitoring temperature data | 28 days
  Proportion of patients able to wear at least one sensor device for ≥50% of days from Day 0 (CAR-T infusion) through Day 28, with ≥12 hours/day of usable data collected (temperature, heart rate).

SECONDARY OUTCOMES:
Feasibility of microsampling | 28 days
  microsample device collects up to 200 microliters (0.04 teaspoons) of blood from the upper arm
Safety of wearable devices | 28 days
  Safety will be measured by skin irritation, rash. Will be assessed using CTCAE criteria version 5 to evaluate by any adverse event definitely, probably or possibly related to the wearable devices
Safety of the microsampling device | 28 days
  Microsampling will be measured by process such as minor bruising, bleeding, or infection. Will be assessed using CTCAE criteria version 5 to evaluate by any adverse event definitely, probably or possibly related to the wearable devices

CONTACTS AND LOCATIONS:
Overall Officials: Surbhi Sidana, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No